CLINICAL TRIAL: NCT06373458
Title: A Single-Center, Two-Arm, Open-Label Phase IIA Clinical Trial to Investigate Efficacy and Safety of Ritlecitinib in Patients With Keloid
Brief Title: Ritlecitinib in Patients With Keloids or Those Undergoing Keloidectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Emma Guttman, Chair, Department of Dermatology, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-01508
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants receiving keloidectomy (Experimental): A total of 20 patients receiving keloidectomy (~50% earlobe keloidectomy cap) at Day 1 as Group 1
  Interventions: Drug: Ritlecitinib
- Participants with no keloidectomy (Experimental): A total of 10 patients with no keloidectomy during the study and with at least one keloid measuring ≥3 cm or multiple keloids, measuring ≥1 cm in length each, as Group 2
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — Ritlecitinib 50mg QD for 36 weeks starting at Day 1

SUMMARY:
Keloids are common, benign cutaneous overgrowths that manifest clinically as raised, hypertrophic, often hyperpigmented lesions which are formed in response to dermal injury or idiopathic stimuli. Although keloids are a common disease, it's exact incidence and prevalence is not known. Despite the debilitating nature of keloids, current treatment modalities are limited in efficacy; there is no universally effective therapy available to patients. The research team hypothesize that ritlecitinib as a JAK3/TEC inhibitor will be able to reverse both the systemic and local keloid disease process by re-establishing immune homeostasis.

DETAILED DESCRIPTION:
This study is a prospective, two-arm, open-label clinical trial to investigate efficacy and safety of ritlecitinib in patients with keloid. The study will take place at Icahn School of Medicine at Mount Sinai. The study will consist of 2 arms: a total of 20 patients receiving keloidectomy and a total of 10 patients with no keloidectomy during the study and with at least one keloid measuring ≥3 cm or multiple keloids, measuring ≥1 cm in length each. Patients will be treated with ritlecitinib 50 mg QD for 36 weeks starting at Day 1. Participants will attend clinic visits at Weeks 2, 4, 8, 12, 20, 28, and 36 for assessments, questionnaires and safety laboratory tests. The follow-up period will be 6 months, with clinic visits at Weeks 48 and 60.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ≥ 18 years of age at the time of signing the informed consent document (not more than 10% of the patients can be > 50 years of age).
* Patient is able to understand and voluntarily sign an informed consent document prior to participation in any study assessments or procedures.
* Patient is able to adhere to the study visit schedule and other protocol requirements.
* Patients who receive keloidectomy at Day 1/ Baseline only (Group 1): Patient has minimum of one keloid measuring ≥2 cm in length on earlobe or ≥3.0 cm in length on areas) other than earlobe, which has failed prior minimally invasive treatments for keloids including topicals and intralesional corticosteroid injections and that can be surgically resected at Day 1/ Baseline.
* Patients who do not receive keloidectomy at Day 1/ Baseline only (Group 2):

  * Patient has a minimum of either one keloid measuring ≥3 cm in length, or multiple keloids, each measuring ≥1 cm in length , which failed prior minimally invasive treatments for keloids including topicals and intralesional corticosteroid injections. However, at least one keloid should not have been treated with surgery, cryotherapy, radiation, or any other procedure that leads to a deformity that interferes with proper clinical assessments.
  * Patient reports either Pain-NRS ≥4 , Itch-NRS ≥4, or DLQI ≥8both at Visit 1 (Screening) and Visit 2 (Baseline)
* Patient is judged to be in otherwise good overall health as judged by the investigator, based on medical history, physical examination, and laboratory testing. (NOTE: The definition of good health means a patient does not have uncontrolled significant co-morbid conditions).
* Ability to take oral medication without crushing, dissolving or chewing tablets.
* Females of childbearing potential (FOCBP) must have a negative pregnancy test at Screening and Day 1/ Baseline. While on ritlecitinib and for at least 28 days after taking the last dose of ritlecitinib, FOCBP who engage in activity in which conception is possible must use the approved contraceptive methods.

Exclusion Criteria:

* Patient has a persistent or recurring bacterial infection requiring systemic antibiotics, or clinically significant viral or fungal or helminth parasitic infections, within 2 weeks of the Screening Visit. Any treatment of such infections must have been completed at least 2 weeks prior to the Screening Visit and no new/recurrent infections should have occurred prior to the Baseline Visit.
* Patient with current or history of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (i.e., Common Variable Immunodeficiency [CVID]), or active or untreated latent tuberculosis.
* Infected with hepatitis B or C virus.
* Patients who have history of single episode of disseminated herpes zoster (HZ) or disseminated herpes simplex or recurrent (> 1 episode of) localized dermatomal HZ
* Patient has clinically significant (as determined by the investigator) renal, hepatic, hematologic, intestinal, endocrine, pulmonary, cardiovascular, neurological, psychiatric, immunologic, or other major uncontrolled diseases that will affect the health of the patient during the study or interfere with the interpretation of study results.
* Patient has a suspected or active lymphoproliferative disorder or malignancy; OR a history of malignancy within 5 years before the Baseline assessment, except for completely treated in situ non-melanoma skin and cervical cancers without evidence of metastasis.
* Any gastrointestinal or metabolic condition that could interfere with the absorption of the oral medication.
* Active alcohol and/or drug abuse.
* History of thrombosis/ thromboembolic event, known coagulopathy.
* Additional skin disease that might interfere with keloid clinical assessments.
* Have hearing loss with progression over the previous 5 years, or sudden hearing loss, or middle or inner ear disease including otitis media, cholesteatoma, Meniere's disease, labyrinthitis, or other auditory condition that is considered acute, fluctuating, or progressive.
* Patient has received a live attenuated vaccine ≤ 30 days prior to study initiation.
* History of adverse systemic or allergic reactions to any component of the study drug.
* Recent surgery excluding keloidectomy within 4 weeks and keloidectomy within 6 months prior to trial initiation.
* Recent cryotherapy within 3 months, laser therapy within 3 months, or radiation or any other procedure within 6 months.
* Use of systemic immunosuppressive medications, including, but not limited to, cyclosporine, systemic or intralesional corticosteroids, mycophenolate mofetil, azathioprine, methotrexate, tacrolimus, or ultraviolet (UV) phototherapy with or without Psoralen Ultraviolet A (PUVA) therapy within 4 weeks prior to trial initiation. Compression garments and silicone sheets may be allowed.
* Treatment with medication that might interfere with blood levels or have a major impact on the clinical readout of the study drug. This includes the following:

  * Patient on concomitant medications that are substrates of CYP3A4 or CYP1A2 with narrow therapeutic index where small concentration changes may lead to serious adverse reactions
  * Patient on concomitant medications that are strong inducers of CYP3A4 as this might cause loss of efficacy of ritlecitinib
* Use of an oral JAK inhibitor (tofacitinib, ruxolitinib, ritlecitinib) within 3 months prior to the Baseline visit.
* Patient has used topical corticosteroids, and/or tacrolimus, and/or pimecrolimus, and/or topical chemotherapy on any keloid lesions within 2 weeks prior to the Baseline visit. These will be allowed during the study on areas other than keloid lesions (if applicable) but not on any keloid lesions.
* Female patient who is pregnant or breast feeding
* FOCBP with unwillingness or inability to use a contraception method during the time of participation in the trial (Appendix 1)
* Abnormality in hematology, chemistry profiles, and ECG during screening:

  * Platelet count: <75000/ mm3
  * Lymphocytes: <600/ mm3
  * Absolute neutrophil count: <1200/ mm3
  * Hemoglobin: <9.0 g/dL
  * ALT or AST: >3.0xULN
  * eGFR: <30 mL/min
  * ECG that demonstrates clinically relevant abnormalities that may affect patient safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence Rate | at 9 months (Visit 9)
  Recurrence Rate at 9 months (Visit 9) in subjects that received keloidectomy
Change in Detroid Keloid Scale Score | Baseline and 9 months (Visit 9)
  Change from Baseline in the Detroit Keloid Scale at 9 months (visit 9) (excluding those without measurable keloids after keloidectomy). Detroit Keloid Scale is a questionnaire consisting of 3 questions that assess the clinical observation (observer keloid assessment) and 4 questions that evaluate the 3 clinical signs of keloids and the impact of keloids on the patient's well-being (patient keloid questionnaire).
  Keloid Severity (Calculated from Total) 0-4 = mild; 5-9 = moderate; 10-14 = severe
  Total scores from 0-14, with higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in Peak keloid tension | Visits 2 (Week 0) and up to visit 11 (Week 60)
  Efficacy of ritlecitinib measured by peak keloid tension. Peak keloid tension measures the "hardness" of the skin using an instrument called a tonometer. Full scale ranges 0-100, with higher scores indicating greater "hardness".
Change in Detroid Keloid Scale Score (DKS) | Visits 2 (Week 0) and up to visit 11 (Week 60)
  Efficacy of Ritlecitnib measured using Detroid Keloid Scale.
  The DKS is a questionnaire consisting of 3 questions that assess the clinical observation (observer keloid assessment) and 4 questions that evaluate the 3 clinical signs of keloids and the impact of keloids on the patient's well-being (patient keloid questionnaire).
  Keloid Severity (Calculated from Total) 0-4 = mild 5-9 = moderate 10-14 = severe
  Total scale from 0-14. Higher scores indicate greater symptom severity.
Change in Pain Numerical Rating Scale (Pain-NRS) | Visits 2 (Week 0) and up to visit 11 (Week 60)
  Efficacy of ritlecitinib measured by Pain-NRS. The NRS will range from 0 (no symptoms) to 10 (severe symptoms). Patients indicate the intensity of pain by choosing a number from 0 (no pain) to 10 (worst imaginable pain) that corresponds to the severity of that symptom, with higher scores indicating higher levels of pain.
Change in Itch-NRS | Visits 2 (Week 0) and up to visit 11 (Week 60)
  Efficacy of ritlecitinib measured by Itch-NRS. The NRS will range from 0 (no symptoms) to 10 (severe symptoms). Patients indicate the intensity of itch by choosing a number from 0 to 10 that corresponds to the severity of that symptom.
  Scale 0-10 0 = No Itch 10 = Worst Itch Imaginable
  Higher scores indicate greater itch severity.
Change in PGIC (Patient Global Impression of Change) | Visits 2 (Week 0) and up to visit 11 (Week 60)
  Efficacy of ritlecitinib measured by Patient Global Impression of Change (PGIC). The PGIC will be used to assess self-reported relieving effect. It will evaluate pain from no change (score 0-1), minimally improved (score 2-3), much improved (score 4-5), and very much improved (score 6-7). Total Scale from 0-87. Higher scores indicate more favorable health outcomes.
  Patients will be asked to choose ONE:
  * No change (or condition has gotten worse) (1)
  * Almost the same, hardly any change at all (2)
  * A little better, but no noticeable change (3)
  * Somewhat better, but the change has not made any real difference (4)
  * Moderately better, and a slight but noticeable change (5)
  * Better and a definite improvement that has made a real and worthwhile difference (6)
  * A great deal better and a considerable improvement that has made all the difference (7)
Change in DLQI (Dermatology Life Quality Index) | Visits 2 (Week 0) and up to visit 11 (Week 60)
  Efficacy of ritlecitinib measured by Dermatology Life Quality Index (DLQI). DLQI is a 10-item questionnaire, each question is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life), thus, higher scores indicate greater impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Results will be provided as aggregated data.